CLINICAL TRIAL: NCT00562991
Title: Monitoring Asthma Treatment Using Exhaled Nitric Oxide
Acronym: NOASTHMA
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Aerocrine AB (Industry)
Responsible Party: Sponsor
Other Study IDs: B30020072436
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2007-11

CONDITIONS: Asthma
Keywords: exhaled NO; asthma; child
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FeNO group: asthma patients, exhaled NO is used to monitor asthma
  Interventions: Device: measurement of exhaled NO is used to guide treatment
- Symptom group: asthma patients, exhaled NO is not used to monitor asthma

INTERVENTIONS:
Device: measurement of exhaled NO is used to guide treatment — exhaled NO
  Groups: FeNO group

SUMMARY:
Asthma is a chronic inflammatory condition in which the airways develop increased responsiveness to various stimuli such as exposure to an allergen, cold air or exercise. It is characterized by airway hyper-responsiveness, inflammation, increased mucus production, and airway obstruction. Since inflammation is an important feature of asthma, the use of non-invasive tests to measure lung inflammation to monitor asthma are of interest.The purpose of the study is to relate costs associated with healthcare utilization and loss of work and school time to the primary health outcome of cumulative number of symptom-free days. This will enable the researchers to determine whether the costs of monitoring exhaled NO to regular management strategy in recently diagnosed asthma will be offset by reductions in other costs of asthma-related care, and, if not, whether the additional costs are likely to be acceptable in terms of the improvement in health outcomes as measured by the additional number of symptom-free days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children, aged 6-14 years
* A documented history of asthma for a period of at least 6 months
* Mild to severe persistent asthma according to GINA guidelines
* A documented history of allergic sensitization (positive skin prick test or specific IgE
* Subject's guardian/parent should be able to complete a symptom score on behalf of the subject.
* Subject's guardian/parent should be able to send a symptom score weekly by sms
* Both parents have to give written informed consent to participate in the study

Exclusion Criteria:

* Received any investigational study medication in the 4 weeks prior to screening Visit
* Significant comorbidity such as concurrent infection, history of prematurity, history of bronchopulmonary dysplasia, cystic fibrosis, other chronic lung diseases, and other severe chronic diseases
* Acute asthma exacerbation within 4 weeks of screening visit
* Hospitalization within 12 weeks of screening visit
* Systemic corticosteroids within 12 weeks of screening visit
* Oral corticosteroid dependence

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: asthmatic children
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2007-10-01 (Actual); Primary Completion 2008-10-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
symptom-free days | 1 year time frame with visits every 3 months

SECONDARY OUTCOMES:
days spent in hospital,emergency room visits,physician or nurse contacts use of drugs, days on which school was missed, number of exacerbations | 1 year time frame

CONTACTS AND LOCATIONS:
Overall Officials: kristine N Desager, PhD, Principal Investigator — University Hospital, Antwerp
Locations (7):
- Belgium (7):
  - University Hospital Antwerp, Antwerp
  - Algemeen Ziekenhuis St Jan, Bruges
  - Univ des enfants Reine Fabiola, Brussels
  - Hôpital Erasme, Brussels
  - Virga Jesseziekenhuis, Hasselt
  - Algemeen ziekenhuis Turnhout, Campus Sint-Jozef, Turnhout
  - CH Peltzer, Verviers

REFERENCES:
- [Derived] Peirsman EJ, Carvelli TJ, Hage PY, Hanssens LS, Pattyn L, Raes MM, Sauer KA, Vermeulen F, Desager KN. Exhaled nitric oxide in childhood allergic asthma management: a randomised controlled trial. Pediatr Pulmonol. 2014 Jul;49(7):624-31. doi: 10.1002/ppul.22873. Epub 2013 Sep 4. PMID 24039119